CLINICAL TRIAL: NCT04275518
Title: A Phase Ib Study to Investigate the Safety, Pharmacokinetics and Pharmacodynamics of APG-115 as a Single Agent or in Combination With Azacitidine or Cytarabine in Patients With Relapse/Refractory AML and Relapsed/Progressed High/Very High Risk MDS
Brief Title: A Phase Ib Study of APG-115 Single Agent or in Combination With Azacitidine or Cytarabine in Patients With AML and MDS.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Collaborators: Suzhou Yasheng Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APG115AC101
Record Dates: First submitted 2020-02-05; First posted 2020-02-19 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Acute Myeloid Leukemia (AML); Myelodysplastic Syndromes (MDS)
Keywords: APG-115; AML; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Azacitidine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APG-115/APG-115+Cytarabine in Relapse/Refractory AML (Experimental)
  Interventions: Drug: APG-115; Drug: Cytarabine
- APG-115/APG-115+Aza in relapsed/progressed high risk MDS (Experimental)
  Interventions: Drug: APG-115; Drug: Azacitidine

INTERVENTIONS:
Drug: APG-115 — APG-115 orally once daily from Days 1 to 7 every 28 days.
Drug: Azacitidine — 75 mg/m^2 SC QD on Days 1- 7 (28-day cycle)
  Arms: APG-115/APG-115+Aza in relapsed/progressed high risk MDS
Drug: Cytarabine — 1g/m^2 IV QD on Days 3-7 (28-day cycle)
  Arms: APG-115/APG-115+Cytarabine in Relapse/Refractory AML

SUMMARY:
Acute myeloid leukemia is a malignant disorder characterized by the rapid, uncontrolled proliferation of malignant clonal hematopoietic stem cells that accumulate as immature, undifferentiated cells (blasts) in the bone marrow and circulation.

APG-115 is a potent and orally active small-molecule MDM2 inhibitor, it binds to MDM2 protein and shows potent cell growth inhibitory activity in vitro with low nanomolar potencies in a subset of human cancer cell lines. APG-115 has demonstrated its strong antitumor activities with either daily or less frequent dosing-schedules in the acute leukemia xenograft models.

This is a phase 1b, open-label, three-stages study that will initially evaluate the safety and PK/PD profile of APG-115 as a single agent, followed by a combination of APG-115 + azacytidine or cytarabine in R/R AML or MDS subjects.

Patients will continue treatment for maximally 6 cycles or until progression of disease or unacceptable toxicity is observed or administrative discontinuation whichever occurs first. Patients who continue to be benefit after 6 cycles' treatment will receive additional cycles of treatment until progression of disease, unacceptable toxicity is observed or administrative discontinuation. (As long as it is proven safe).

DETAILED DESCRIPTION:
Stage 1: This will be a 3+3 dose escalation to determine the DLTs and MTD/RP2D of APG-115 given according to the different dose levels once daily from Days 1 to 7 every 28 days.

Stage 2: After stage 1 of APG-115 single agent dose escalation first cycle is completed, stage 2 can be initiated with the combination regimen. This will be a 3+3 dose escalation to determine the MTD/RP2D and DLTs of APG-115 + AZA(arm A)/Cytarabine (arm B)combination.

Stage 3: dose expansion of the combination regimes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of histologically confirmed relapsed or refractory (R/R) acute myeloid leukemia by WHO classification or relapsed/progressed high/very high risk MDS (score≥4.5) according to IPSS-R risk stratification
2. Age >/= 18 years.
3. Adequate organ function
4. Subject must have a projected life expectancy of at least 12 weeks.
5. ECOG performance status of 0-1.
6. Patient must have the ability to understand the requirements of the study and signed informed consent. A signed informed consent by the patient or his legally authorized representative is required prior to their enrollment on the protocol.
7. Subject has a white blood cell count< 50 × 109/L. Note: Hydroxyurea is permitted to meet this criterion.

Exclusion Criteria:

1. Subject has acute promyelocytic leukemia.
2. Patients must not have had leukemia biotherapy 4 weeks prior to starting investigational drug, or less than 5 half-lives small molecular targeted drug therapy, or 28 days any anti-cancer therapy (whichever is longer)
3. Uncontrolled intercurrent illness including, but not limited to active uncontrolled infection, symptomatic congestive heart failure (NYHA Class III or IV), unstable angina pectoris, clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
4. Active infection requiring systemic antibiotic/antifungal medication, known clinically active hepatitis B or C, or HIV infection.
5. Participants who have received allogeneic HSCT, or autologous HSCT within 12 months.
6. Patients with active, uncontrolled CNS leukemia will not be eligible.
7. Any prior systemic MDM2-p53 inhibitor treatment
8. Any other condition or circumstance that would, in the opinion of the investigator, make the patient unsuitable for participation in the study.
9. Subject has a history of other malignancies within 2 years prior to study entry, with the exception of:

   * Adequately treated in situ carcinoma of the cervix uteri or carcinoma in situ of breast;
   * Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin;
   * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intention: requires discussion with sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2020-07-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | From day 1 to the end of cycle 1 (each cycle is 28 days).
  DLT will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE, version 5) by organ system. DLT will be defined as clinically significant drug-related adverse events during the Cycle one.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Evaluated for response by the end of cycle 1 and cycle 2, and then 2 months thereafter till complete 6 cycles treatment or 1 month after last dose (each cycle is 28 days).
  ORR is defined by CR + CRi+ PR (according to IWG AML（2003）and IWG MDS（2006）criteria)
Overall survival (OS) | Measured up to 6 months after the last subject has received treatment.
  From date of treatment start until the date of death due to any cause or date of termination of the study, whichever came first. Termination of the Study: The last subject has completed at least 6 cycle's treatment or the subject discontinues treatment for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, M.D., Principal Investigator — Blood Diseases Hospital Chinese Academy of Medical Sciences
Locations (14):
- China (14):
  - The First Hospital of Peking University, Beijing, Beijing Municipality
  - Guangzhou panyu central hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Henan Provincial Oncology Hospital, Zhengzhou, Henan
  - Union Hospital medical college Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The First Affilated Hospital of Ganzhou Medical University, Suzhou, Jiangsu
  - The First affiliated hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - First Hospital of Jilin University, Changchun, Jilin
  - Shanghai Jiao Tong University school of medicine Ruijing Hospital, Shanghai, Shanghai Municipality
  - Shanghai Sixth people's Hospital, Shanghai, Shanghai Municipality
  - Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality